CLINICAL TRIAL: NCT03436368
Title: Continuous Spinal Anesthesia for Renal Transplant Recipients
Brief Title: Continuous Spinal Anesthesia in Renal Transplantation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CSARTR60
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Renal Failure Chronic; Transplant;Failure,Kidney; Anesthesia
Keywords: Continuous spinal anesthesia; General anesthesia; Renal transplantation; Chronic renal failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Using computer & sealed envelope randomization, patients are assigned to receive either continuous spinal anesthesia [CSA group: n =30] or general anesthesia [GA group: n=30]
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSA group (Active Comparator): Continuous Spinal Anesthesia
  Interventions: Procedure: Continuous spinal anesthesia
- GA group (Active Comparator): General Anesthesia
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Continuous spinal anesthesia — Continuous spinal anesthesia will be performed for patients of the CSA group at the L3-L4 intervertebral space using Spinocath (B. Braun, Melsungen, Germany). After the cerebrospinal fluid is aspirated, 7.5 mg hyperbaric Bupivacaine 0.5% (1.5 ml) together with 25 micrograms Fentanyl (0.5 ml) will be injected intra-thecally. Supplemental injections will be given in aliquots of 5 mg hyperbaric Bupivacaine 0.5% (1 ml) if the sensory block is lower or reseeds, during surgery, below T6 dermatome.
  Arms: CSA group
Procedure: General anesthesia — Anesthesia will be induced with intra-venous administration of Fentanyl (2 micrograms/kg), Ptopofol (1-2 mg/kg) and Atracurium (0.5 mg/kg). Maintenance will be achieved with 0.8-1.5% Isoflurane in an O2 / air mixture, an Atracurium infusion at 0.5 mg/kg/hr and a Fentanyl infusion at 1 micrograms/kg/hr.
  Arms: GA group

SUMMARY:
Renal transplantation is now recognized as a treatment of choice for patients with end-stage renal disease. An adequate anesthetic technique should achieve hemodynamic stability and enhance perfusion of the transplanted kidney. The aim of this study is to assess the use & effects of continuous spinal anesthesia for kidney transplantation recipients, compared with balanced general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA class III or IV
* End-stage renal disease
* Renal transplantation candidate patients

Exclusion Criteria:

* Any condition contra-indicating regional anesthesia
* Coagulopathy
* Allergic to any of the drugs used during the procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean ABP | 12 hours
  Change in Mean Arterial Blood Pressure measured in mmHg.

SECONDARY OUTCOMES:
Visual Analogue Score for pain "VAS" | 12 hours
  Visual Analogue Score for pain measures the degree of pain experienced by the patient during the procedure. VAS is graded from 0-10 [where 0=no pain, 10= worst pain].
Patient satisfaction score | 24 hours
  Patient satisfaction Score defines the degree of patient satisfaction with the anesthetic experience and is assessed after recovery. It is graded as excellent "E" (best score), fair "F" or poor "P" (worst score).

CONTACTS AND LOCATIONS:
Overall Officials: Nazmy E Seif, MD, Study Chair — Kasr Al-Ainy Hospital, Cairo University
Locations (1):
- Kasr Al-Ainy Hospital, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided